CLINICAL TRIAL: NCT02075307
Title: Highbush Blueberries, the DNA-damage of Obesity, Somatic Mutations and Metabolic Syndrome
Brief Title: Effect of Blueberry Consumption on Metabolic Syndrome & DNA Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: U.S. Highbush Blueberry Council (Other); USDA Agricultural Research Station in Albany, CA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-033
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Metabolic Syndrome; Insulin Resistance; DNA Damage
Keywords: insulin; diabetes; obesity; DNA damage; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry Powder (Experimental): The intervention group will receive the Blueberry freeze-dried powder equivalent to 1 cup of whole Blueberries twice a day for 8 weeks (i.e. 2 cups/day).
  Interventions: Dietary Supplement: Blueberry Powder
- Placebo Powder (Placebo Comparator): The placebo group will receive placebo powder in the same amounts for the same duration.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blueberry Powder
  Arms: Blueberry Powder
Dietary Supplement: Placebo
  Arms: Placebo Powder

SUMMARY:
Obesity usually brings with it disturbances in the body that increase the chances of developing serious diseases like diabetes and cancer. These disturbances include one or more symptoms of a condition called "metabolic syndrome" that often leads to diabetes. High levels of damage to the DNA that makes up our chromosomes have also been observed in obese people. It is possible that these two disturbances are connected. The goal of this project is to test this whether consumption of blueberries will improve these abnormalities.

DETAILED DESCRIPTION:
Unbalanced diets rich in refined carbohydrate calories, saturated fats, and trans fats, but low in vitamins, minerals, fiber, polyphenolics and ω-3 fatty acids are common in the United States, particularly among the obese. Insulin resistance and high levels of DNA damage commonly accompany obesity. There also appears to be a relationship between oxidative DNA-damage and biomarkers that characterize metabolic syndrome. The bioactivity of blueberries is usually attributed to their high content of polyphenolics which can reduce oxidative DNA damage. Since oxidative damage to mitochondrial DNA is a suggested causal factor leading to increased insulin resistance, we will test if blueberry consumption can be an ameliorative dietary factor for insulin resistance as well. If blueberry consumption both shifts metabolism away from insulin resistance and reduces DNA damage, it may be a useful tool to assist in understanding relationships between these two obesity-associated conditions.

ELIGIBILITY:
Inclusion criteria:

1. Age 30-60 years;
2. BMI > 30;
3. Blood pressure <140/90 mmHg without antihypertensive medicines or with a stable dose of antihypertensive medicines (no change in last 3 months).;
4. Insulin resistance (HOMA/IR) > 2.0;
5. Willing to restrict intake of high polyphenol-containing foods during the trial period;
6. Willing to forego intake of nutritional supplements other than a multivitamin;
7. Willing to maintain their current daily level of exercise throughout the study.

Exclusion criteria:

1. Known diabetes mellitus according to the 2013 ADA criteria;
2. Medications known to affect glucose metabolism;
3. Weight loss pharmacotherapy;
4. Lipid-lowering medication;
5. Untreated thyroid or chronic liver, renal, or cardiovascular disease;
6. Smoking;
7. Pregnancy- a negative urine pregnancy test will be documented for any women participants of childbearing age prior to enrollment.
8. History of allergic reactions to blueberries.
9. Any pathological condition known to alter white blood cell count over the previous 6 months;
10. Exposure to drugs known to cause mutations or radiation within the previous 6 months;
11. Alcohol consumption greater than 2 drinks/d for males and 1 drink/d for females.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-01; Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
DNA damage in peripheral blood mononuclear cells | Baseline and 2 months
  DNA double-stranded breaks (DSBs) will be measured.

SECONDARY OUTCOMES:
Insulin resistance | Baseline and 2 months
  Insulin resistance will be measured by a 2-hr glucose tolerance test.

OTHER OUTCOMES:
Thiol/Redox changes | Baseline and 2 months
  Metabolomic profile measuring shifts in the plasma redox environment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ames, PhD, Principal Investigator — Children's Hospital & Research Center at Oakland; Ashutosh Lal, MD, Principal Investigator — Children's Hospital & Research Center at Oakland
Locations (1):
- Children's Hospital & Research Center Oakland, Oakland, California, United States